CLINICAL TRIAL: NCT06770881
Title: Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Antitumor Activity of JSKN033 in Chinese Subjects with Advanced Malignant Tumors
Brief Title: JSKN033 in Chinese Subjects with Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSKN033-102
Record Dates: First submitted 2024-12-27; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JSKN033 (Experimental)
  Interventions: Drug: JSKN033

INTERVENTIONS:
Drug: JSKN033 — JSKN033 should be administered subcutaneously on the first day of each week cycle/ each 2-week cycle

SUMMARY:
This is a phase I/II multicenter study to evaluate the safety and efficacy of JSKN033 in Chinese subjects with unresectable locally advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand informed consent form, voluntarily participate and sign informed consent form.
2. Age ≥18 year (at the time consent is obtained), male or female.
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Has a Life expectancy ≥3 months.
5. Has a pathologically documented advanced/unresectable or metastatic solid malignant tumor that is refractory to or intolerable with standard treatment.
6. Has at least 1 measurable lesion at baseline according to RECIST 1.1 criteria.
7. Must have adequate organ function prior to the start of JSKN033.
8. Negative urine/serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner.

Exclusion Criteria:

1. Has clinically active brain metastases.
2. Previously received any other investigational drug within 28 days prior to enrollment.
3. Previously received local palliative treatment within 14 days prior to enrollment.
4. Previously received major surgeries within 28 days prior to enrollment.
5. Need to receive continuous administration of corticosteroids or immunosuppressants for 7 days within 14 days prior to enrollment.
6. Previously received live vaccine within 28 days prior to enrollment.
7. Previously received antibody conjugate drug with topoisomerase I inhibitor.
8. Has a history of other primary malignant tumors within 5 years prior to enrollment.
9. Has uncontrolled comorbidities as specified by the protocol.
10. Has a history of interstitial pneumonia/lung disease requiring systemic hormonal therapy, or suspected interstitial pneumonia/lung disease that cannot be ruled out by imaging during screening period.
11. Subjects with uncontrolled large serous cavity effusion or moderate to large serous cavity effusion requiring repeated drainage (recurrent within 2 weeks after intervention) such as pleural effusion, pericardial effusion, ascites, etc.
12. Toxicities of previous antitumor therapy did not resolve to grade 1 defined by CTCAE v5.0.
13. Has a history of life-threatening anaphylaxis or known hypersensitivity to any component or excipient to the study drug.
14. Has a history of allogeneic bone marrow or organ transplantation.
15. Pregnant or breastfeeding female patients.
16. Other conditions that the investigator considers unsuitable to participate in this clinical trial, including but not limited to psychiatric disorders, alcoholism or drug abuse, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 12 months
  Incidence of DLT in the dose escalation period.
Maximum Tolerated Dose (MTD) or recommend Phase II dose (RP2D). | Up to 12 months
  Based on safety and efficacy data.
Percentage of Participants Experiencing Any Treatment Emergent Adverse Events (TEAE) and Treatment Related Adverse Events (TRAE) | Throughout the duration of the study, approximately 2 years
  TEAE and TRAE were graded according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

SECONDARY OUTCOMES:
Anti-drug antibodies (ADA) and neutralizing antibodies | Throughout the duration of the study, about 2 years
  Status (positive or negative) and serum titers of anti-JSKN033 antibody.
Objective response rate (ORR) | Throughout the duration of the study, about 2 years
  ORR is determined by investigators based on RECIST 1.1 criteria.
Disease control rate (DCR) | Throughout the duration of the study, about 2 years
  DCR is determined by investigators based on RECIST 1.1 criteria.
Progression-free survival (PFS) | Throughout the duration of the study, about 2 years
  PFS is defined as the time from the date of the first dose to the earlier of the dates of the first objective documentation of radiographic disease progression or death due to any cause.
Maximum concentration (Cmax) | Throughout the duration of the study, about 2 years
  Categories: JSKN003, total antibody (Tab) , payload of JSKN003 and envafolimab.
Time at which Cmax is reached (Tmax) | Throughout the duration of the study, about 2 years
  Categories: JSKN003, total antibody (Tab) , payload of JSKN003 and envafolimab.
Area under the drug concentration-time curve (AUC) to the last observable concentration (AUClast) | Throughout the duration of the study, about 2 years
  Categories: JSKN003, total antibody (Tab) , payload of JSKN003 and envafolimab.

CONTACTS AND LOCATIONS:
Overall Officials: XiaoHua Wu, MD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No